CLINICAL TRIAL: NCT02086890
Title: Modulating Ocular/Retinal Blood Flow and Visual Function in Retinitis Pigmentosa
Brief Title: Electro-acupuncture and Transcorneal Electrical Stimulation (TES) for Retinitis Pigmentosa
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Kenneth Seger, Associate Professor, HPD-College of Optometry, Nova Southeastern University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01311402F; R21EY023720 (NIH)
Record Dates: First submitted 2014-03-10; First posted 2014-03-13 (Estimated); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Retinitis Pigmentosa
Keywords: retinitis pigmentosa; acupuncture; electroacupuncture; transcorneal electrical stimulation; microcurrent
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Electro-acupuncture (Experimental): Electro-acupuncture applied to acupoints around the eye and traditional needle acupuncture applied to acupoints throughout the body at 10 half-hour sessions over 2 weeks
  Interventions: Device: Electro-acupuncture
- Sham Electro-acupuncture (Sham Comparator): No electro-acupuncture applied to non-acupoints around the eye and traditional needle acupuncture applied to non-acupoints throughout the body; i.e., to locations not on the acupuncture meridians; at 10 half-hour sessions over 2 weeks
  Interventions: Device: Sham Electro-acupuncture
- Laser acupuncture (Experimental): Laser applied to acupoints throughout the body at 10 sessions each lasting 15 minutes over a 2 week period
  Interventions: Device: Laser Acupuncture
- Sham Laser acupuncture (Sham Comparator): An inactive sham laser (red light only) applied to non-acupoints throughout the body; i.e., to locations not on the acupuncture meridians; at 10 sessions each lasting 15 minutes over a 2 week period
  Interventions: Device: Sham laser acupuncture
- Transcorneal Electrical Stimulation (Experimental): Transcorneal Electrical Stimulation at 150% individual phosphene threshold applied to both eyes using DTL electrodes at 6 weekly 30 minute sessions
  Interventions: Device: Transcorneal Electrical Stimulation
- Sham Transcorneal Electrical Stimulation (Sham Comparator): Sham Transcorneal Electrical Stimulation at 0% individual phosphene threshold (no stimulation) applied to both eyes using DTL electrodes at 6 weekly 30 minute sessions
  Interventions: Device: Sham transcorneal electrical stimulation

INTERVENTIONS:
Device: Electro-acupuncture
  Arms: Electro-acupuncture
Device: Laser Acupuncture
  Arms: Laser acupuncture
Device: Transcorneal Electrical Stimulation
  Arms: Transcorneal Electrical Stimulation
Device: Sham Electro-acupuncture
  Arms: Sham Electro-acupuncture
Device: Sham laser acupuncture
  Arms: Sham Laser acupuncture
Device: Sham transcorneal electrical stimulation
  Arms: Sham Transcorneal Electrical Stimulation

SUMMARY:
Measures of vision in RP patients receiving promising therapy using transcorneal electrical stimulation.

DETAILED DESCRIPTION:
Retinitis pigmentosa (RP) is a slowly progressive retinal degeneration for which there is no proven treatment. Patients are interested in trying alternative therapies to try to reduce their vision loss, but only limited research evidence exists to support their use and potential benefit. The goal of this research project is to gain a better understanding of possible changes in ocular and retinal blood flow and measures of vision in RP patients receiving two promising therapies, electroacupuncture and transcorneal electrical stimulation. We are currently only doing transcorneal electrical stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Diagnosis of retinitis pigmentosa (RP)
* Best-corrected visual acuity better than 20/400 in at least one eye
* More than 20% loss of Goldmann Visual Field area (III4e test target) in at least one eye
* Able and willing to participate in all study visits for a ~4-6 month period
* Provide informed consent

Exclusion Criteria:

* Very severe vision losses in both eyes (e.g., hand motions or light perception only) with difficulty performing the proposed vision tests
* Vision loss due to ocular diseases other than RP, cystoid macular edema, or cataracts
* Schedules do not permit participation in all study visits
* Previous acupuncture or TES treatment for RP
* Inability to understand study procedures or communicate responses to visual stimuli in a consistent manner (cognitive impairment)
* Dementia; Long or short-term memory loss
* Unable to read or speak English
* Smoking, excessive alcohol, or illegal drug use
* Receiving current psychiatric care (i.e. unstable emotional and mental health status)
* History of excessive bleeding
* Reduced general health and/or systemic medications that may diminish the potential response to the electroacupuncture treatments
* Implanted cardiac pacemaker
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Significant changes from baseline in Goldmann visual field area in both eyes | twice at baseline, then 2 weeks, 6 weeks and 12 weeks post-intervention initiation
  Using Haig-Streit Octopus perimeter

SECONDARY OUTCOMES:
Significant changes from baseline in best-corrected ETDRS visual acuity at both 2 weeks and 6 weeks post-intervention initiation | twice at baseline, then 2 weeks, 6 weeks and 12 weeks post-intervention initiation
  Using Pelli-Robson visual acuity charts
Changes in Macular edema Optical Coherence Tomography (OCT) | twice at baseline, then 2 weeks, 6 weeks and 12 weeks post-intervention initiation
  Using Optical Coherence Tomography
Significant changes from baseline in contrast sensitivity at both 2 weeks and 6 weeks post-intervention initiation | twice at baseline, then 2 weeks, 6 weeks and 12 weeks post-intervention initiation
  Using Adaptive Sensory Technology Quick CSF
Significant changes from baseline in Dark adaptation function at both 2 weeks and 6 weeks post-intervention initiation | twice at baseline, then 2 weeks, 6 weeks and 12 weeks post-intervention initiation
  Using the AdaptDx by Maculogix

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth R Seger, OD, MSc, Principal Investigator — Faculty
Locations (1):
- Nova Southeastern University; College of Optometry, Fort Lauderdale, Florida, United States

REFERENCES:
- [Background] Bittner AK, Gould JM, Rosenfarb A, Rozanski C, Dagnelie G. A pilot study of an acupuncture protocol to improve visual function in retinitis pigmentosa patients. Clin Exp Optom. 2014 May;97(3):240-7. doi: 10.1111/cxo.12117. Epub 2013 Oct 29. PMID 24773463
- [Result] Bittner AK, Seger K. Longevity of visual improvements following transcorneal electrical stimulation and efficacy of retreatment in three individuals with retinitis pigmentosa. Graefes Arch Clin Exp Ophthalmol. 2018 Feb;256(2):299-306. doi: 10.1007/s00417-017-3858-8. Epub 2017 Dec 8. PMID 29222719
- [Result] Bittner AK, Seger K, Salveson R, Kayser S, Morrison N, Vargas P, Mendelsohn D, Han J, Bi H, Dagnelie G, Benavente A, Ramella-Roman J. Randomized controlled trial of electro-stimulation therapies to modulate retinal blood flow and visual function in retinitis pigmentosa. Acta Ophthalmol. 2018 May;96(3):e366-e376. doi: 10.1111/aos.13581. Epub 2017 Nov 11. PMID 29130647
- [Result] Kayser S, Vargas P, Mendelsohn D, Han J, Bi H, Benavente A, Bittner AK. Reduced Central Retinal Artery Blood Flow Is Related to Impaired Central Visual Function in Retinitis Pigmentosa Patients. Curr Eye Res. 2017 Nov;42(11):1503-1510. doi: 10.1080/02713683.2017.1338350. Epub 2017 Sep 14. PMID 28910168